CLINICAL TRIAL: NCT02315872
Title: The Effect of ACTH (Acthar) on Measures of Chronic Fatigue in Patients With Relapsing Multiple Sclerosis.
Brief Title: ACTH for Fatigue in Multiple Sclerosis Patients
Acronym: ACTH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Providence Health & Services (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13-120A
Record Dates: First submitted 2014-12-09; First posted 2014-12-12 (Estimated); Results first posted 2019-08-13 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-08

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Multiple Sclerosis; Acthar Gel; ACTH; Fatigue
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis; Fatigue | interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ACTH (Experimental): The study drug (ACTH 40 units) will be given subcutaneously twice weekly for 2 weeks. If the patient tolerates this dosage regimen, the dose will be increased to 80 units twice weekly. If the 80 unit dosage is not tolerated, the dosage will be reduced to 40 units twice weekly for the remainder of the 24 week participation. The weekly doses will be given 3 days apart, for example, on every Monday and Thursday or every Tuesday and Friday.
  Interventions: Drug: ACTH
- Placebo (Placebo Comparator): Placebo will be given subcutaneously twice weekly for 28 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ACTH — ACTH injections twice weekly for 28 weeks.
  Other Names: Acthar Gel; Repository Corticotropin Injection
  Arms: ACTH
Drug: Placebo — Placebo injections twice weekly for 28 weeks.
  Other Names: Control
  Arms: Placebo

SUMMARY:
This is a study of Acthar gel (ACTH) in patients with relapsing multiple sclerosis who are experiencing chronic fatigue.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, placebo-controlled study to demonstrate the safety, tolerability, and effect of ACTH on fatigue in patients with relapsing multiple sclerosis (RMS). The primary objective of this study is to assess the efficacy of ACTH versus placebo in reducing fatigability in patients with RMS. Secondary objectives include assessment of the tolerability and safety of twice-weekly ACTH treatment vs. placebo and evaluation of ACTH on depression, sleepiness, and quality of life measures and correlations between these measures.

ELIGIBILITY:
Inclusion Criteria:

* Have documented diagnosis of Relapsing MS as defined by McDonald Criteria 2011 Revision for at least 6 months
* Have been treated with interferon beta 1a or 1b, glatiramer acetate, fingolimod, dimethyl fumarate, or teriflunomide for at least 6 months, with reported adherence rate of at least 75%, at time of screening
* Have an Kurtzke Expanded Disability Status Scale (EDSS) score of 0 to 4, inclusive
* Have Modified Fatigue Impact Scale (MFIS) ≥ 38 or Functional Systems Scores (FSS) ≥ 36, Beck Depression Inventory-II (BDI-II) greater than or equal to 19, and Expanded Disability Status Scale (EDSS) greater than or equal to 9
* Women of childbearing potential must employ proven methods to prevent pregnancy during the course of the trial
* Able to understand the purpose and risks of the study
* Must be willing to sign an inform consent
* Must be willing to follow the protocol requirements
* Subject must agree not to receive any live or live-attenuated vaccine during the trial

Exclusion Criteria:

* Have any of the contraindications for Acthar Gel as listed in the approved label, including sensitivity to proteins of porcine origin.
* Had treatment of systemic or oral corticosteroids of any type in 90 days prior to baseline/randomization
* Had a relapse or documented objective neurologic worsening in 90 days prior to baseline/randomization
* Has concurrent neurological disease other than multiple sclerosis
* History of sleep apnea
* History (within 90 days) of nocturnal pain and / or nocturnal spasms that interferes with or disrupts sleep, or uncontrolled nocturnal restless leg syndrome
* History of psychosis, bipolar disorder, mania/hypomania
* History of coronary heart disease, congestive heart failure, chronic pulmonary disease, emphysema, anemia, bleeding disorder, gastrointestinal bleeding, intestinal ulcer, clinically significant cardiac arrhythmia, Type I or II diabetes, uncontrolled hypertension, seizure disorder, cardiac arrhythmia, immune deficiency disorder, HIV-AIDS, tuberculosis, or dysthyroidal state (patients with a history of hypothyroidism or hyperthyroidism, which has been corrected to physiological levels will not be excluded)
* History of substance abuse, other than tobacco within the past 5 years or current alcohol dependence
* Current use of cannabis, opiates, benzodiazepines, barbiturates, gabapentin, pregabalin, topiramate, divalproex sodium, carbamazepine, oxcarbazepine, or any gaba-ergic medications other than tizanidine or Baclofen, which are permitted for spasticity treatment
* History of any malignant neoplasm except for past basal cell or squamous cell carcinoma of the skin, that has been successfully treated prior to the screening visit
* History of psychosis or history of use of neuroleptics including, but not restricted to, haloperidol, chlorpromazine, aripiprazole, olanzapine, risperidone
* History of suicide attempt, current suicidal thinking or is preparing for suicide
* Current use of Amphetamines or methylphenidate
* Current use of modafinil, or armodafinil
* Current use of amantidine
* The subject must have had a medication-free interval of:

  a. 7 days for prior use of: i. methylphenidate, amphetamine or dextroamphetamine ii. modafinil or armodafinil iii. diphenhydramine, phenylephrine, loratadine iv. gabapentin, pregabalin, topiramate, valproate/divalproex v. oxcarbazepine vi. codeine, hydrocodone, oxycodone, diphenhydramine, phenylephrine, gabapentin, pregabalin, topiramate, valproate/divalproex, oxcarbazepine, codeine, hydrocodone, oxycodone b. 14 days for prior use of: i. desloratadine ii. Amantidine iii. alprazolam, lorazepam, morphine, hydromorphone, amantidine, alprazolam, lorazepam iv. morphine, hydromorphone c. 28 days for prior use of: i. clonazepam ii. cannabis or other cannabinoids d. 90 days for prior use of carbamazepine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-05-22 (Actual); Primary Completion 2017-06-20 (Actual); Study Completion 2018-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanely Cohan, MD, PhD, Principal Investigator — Providence Health & Services
Locations (5):
- United States (5):
  - North Central Neurology Associates, PC, Cullman, Alabama
  - Providence Medical Group - Medford Neurology, Medford, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Swedish Medical Center, Seattle, Washington
  - MultiCare Health System -- Institute for Research and Innovation, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Providence Health & Services Brain and Spine Institute — http://oregon.providence.org/our-services/p/providence-brain-and-spine-institute/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ACTH | Placebo
Started | 4 | 4
Completed | 1 | 3
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ACTH | Placebo | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 7
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Full Range); unit: years] | 54.5 [45 to 65] | 52 [30 to 67] | 53.25 [30 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 3 | 4 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 8
Modified Fatigue Impact Scale (MFIS) [Mean (Full Range); unit: units on a scale] — This instrument provides an assessment of the effects of fatigue in terms of physical, cognitive, and psychosocial functioning. The full-length MFIS consists of 21 items scored as units on a scale between 0-84. A higher score on the MFIS indicates a greater impact of fatigue on a patient's activities.
  units on a scale | 47.75 [38 to 58] | 48.5 [39 to 71] | 48.125 [38 to 71]
Fatigue Severity Scale [Mean (Full Range); unit: units on a scale] — The Fatigue Severity Scale is a 9-item scale which measures the severity of fatigue and its effect on a person's activities and lifestyle in patients with a variety of disorders as units on a scale between 9-63. Higher scores indicate a greater severity of fatigue.
  units on a scale | 53.25 [45 to 56] | 44.5 [37 to 57] | 48.875 [37 to 57]
Beck Depression Inventory-II (BDI-II) [Mean (Full Range); unit: units on a scale] — The BDI-II is a 21-item self-report multiple-choice inventory used as an indicator of the severity of depression. Scoring is measured with units on a scale between 0-63. A higher score indicates a greater severity of depression.
  units on a scale | 13 [7 to 19] | 9.75 [4 to 16] | 11.375 [4 to 19]
The Epworth Sleepiness Scale (ESS) [Mean (Full Range); unit: units on a scale] — The ESS is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3), their usual chances of dozing off or falling asleep while engaged in eight different activities. The ESS score (the sum of 8 item scores, 0-3) can range from 0 to 24. The higher the ESS score, the higher that person's average sleep propensity in daily life, or their 'daytime sleepiness'.
  units on a scale | 7 [3 to 9] | 10.75 [2 to 19] | 8.875 [2 to 19]
Short Form (36) Health Survey (SF-36) Mental Score [Mean (Full Range); unit: units on a scale] — The SF-36 is a 36-item, patient-reported survey of patient health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability.
  units on a scale | 43 [36 to 57] | 47.5 [37 to 55] | 45.25 [36 to 57]
SF-36 Physical Score [Mean (Full Range); unit: units on a scale] — Measure Description: The SF-36 is a 36-item, patient-reported survey of patient health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability.
  units on a scale | 37.75 [33 to 44] | 45 [32 to 56] | 41.25 [33 to 56]

OUTCOME MEASURES:

1. Primary Outcome: Fatigue at 28 Weeks
Description: Patient-reported levels of fatigue as measured by score on the Modified Fatigue Impact Scale (MFIS) and the Fatigue Severity Scale (FSS) at 28 weeks. The full-length MFIS consists of 21 items. A higher score on the MFIS indicates a greater impact of fatigue on a patient's activities. The FSS is a 9-item scale which measures the severity of fatigue and its effect on a person's activities and lifestyle in patients with a variety of disorders. Higher scores on each scale indicate a greater severity of fatigue.
Time Frame: 28 weeks
Measure: Median (Full Range); unit: score on a scale
Arm/Group | ACTH | Placebo
Number analyzed (Participants) | 4 | 4
score on a scale
  MFIS | 56.50 [21 to 74] | 29.00 [5 to 74]
  FSS | 55.00 [25 to 63] | 40.00 [25 to 57]

2. Secondary Outcome: Depression at 28 Weeks
Description: Patient-reported depression as measured by the Beck Depression Inventory-II (BDI-II) at 28 weeks. The BDI-II is a 21-item self-report multiple-choice inventory used as an indicator of the severity of depression. A higher score indicates a greater severity of depression.
Time Frame: 28 weeks
Measure: Median (Full Range); unit: score on a scale
Arm/Group | ACTH | Placebo
Number analyzed (Participants) | 4 | 4
score on a scale | 16.50 [0 to 22] | 40.00 [25 to 57]

3. Secondary Outcome: Sleepiness at 28 Weeks
Description: Patient-reported daytime sleepiness as measure by the Epworth Sleepiness Scale (ESS) at 28 weeks. The ESS is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3), their usual chances of dozing off or falling asleep while engaged in eight different activities. The ESS score (the sum of 8 item scores, 0-3) can range from 0 to 24. The higher the ESS score, the higher that person's average sleep propensity in daily life, or their 'daytime sleepiness'.
Time Frame: 28 weeks
Measure: Median (Full Range); unit: score on a scale
Arm/Group | ACTH | Placebo
Number analyzed (Participants) | 4 | 4
score on a scale | 11.00 [2 to 16] | 7.00 [1 to 19]

4. Secondary Outcome: Quality of Life at 28 Weeks
Description: Patient-reported quality of life as measured by the 36-Item Short Form Health Survey (SF-36) at 28 weeks. The SF-36 is a 36-item, patient-reported survey of patient mental and physical health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability.
Time Frame: 28 weeks
Measure: Median (Full Range); unit: score on a scale
Arm/Group | ACTH | Placebo
Number analyzed (Participants) | 4 | 4
score on a scale
  SF-36 Mental | 39.50 [25 to 57] | 49.00 [34 to 68]
  SF-36 Physical | 37.50 [30 to 57] | 45.00 [30 to 57]

ADVERSE EVENTS:
Time Frame: Data was collected over 28 weeks.
Arm/Group | ACTH | Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 4/4 | 3/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACTH (N=4) | Placebo (N=4)
bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Sinus infection (Infections and infestations) | 1 (1) | 1 (1)
Flu (Infections and infestations) | 2 (2) | 0 (0)
incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1)
heartburn (Gastrointestinal disorders) | 0 (0) | 1 (1)
insomnia (General disorders) | 1 (1) | 1 (1)
agitation (General disorders) | 1 (1) | 0 (0)
anxiety (General disorders) | 1 (1) | 0 (0)
depression (General disorders) | 1 (1) | 1 (1)
fatigue (General disorders) | 1 (1) | 0 (0)
confusion (General disorders) | 1 (1) | 0 (0) — difficulty word finding
memory loss (General disorders) | 1 (1) | 0 (0)
irritability (General disorders) | 1 (1) | 0 (0)
injection site reaction (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (3)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0)
Yeast infection (Infections and infestations) | 0 (0) | 1 (1)
worsening vision (Eye disorders) | 0 (0) | 1 (1) — worsening vision due to cataract
pain (General disorders) | 0 (0) | 1 (5) — wrist,elbow, rib, toe, and knee pain related to a fall
weight gain (General disorders) | 0 (0) | 1 (1)
worsening asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
weakness (General disorders) | 1 (1) | 1 (1) — right leg weakness
loss of coordination (General disorders) | 0 (0) | 1 (1) — right hand
Worsening muscle spasticity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Left shoulder
Broken toe (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Left pinkie toe
weight gain (General disorders) | 2 (2) | 0 (0)
decreased cutaneous sensation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — feet
dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
plantar dysthesia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
systolic aortic murmur (Cardiac disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 1 (1) | 0 (0)
edema (General disorders) | 1 (1) | 0 (0) — pitting, lower limbs
diaphoresis (General disorders) | 1 (1) | 0 (0)
syncope (General disorders) | 1 (1) | 0 (0)
hypertension (Cardiac disorders) | 1 (1) | 0 (0)
pain and numbness (General disorders) | 0 (0) | 1 (1) — Left hip and arm
enlarged prostate (Renal and urinary disorders) | 1 (1) | 0 (0)
appendicitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
colonic diverticula (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-30): https://cdn.clinicaltrials.gov/large-docs/72/NCT02315872/Prot_SAP_000.pdf